CLINICAL TRIAL: NCT07032454
Title: Investigation of Hand Reaction Speed and Manual Dexterity in Young Adults With Caffeine Dependence
Brief Title: Hand Reaction Speed and Manual Dexterity & Caffeine Dependence
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Assoc.Prof.Dr., PhD, Saglik Bilimleri Universitesi
Other Study IDs: Caffeine_1
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Caffeine Group (≥300 mg/day): Individuals consuming 300 mg or more of caffeine daily, meeting DSM-5/ICD-10 criteria for caffeine dependence.
  Interventions: Other: High Caffeine Consumption
- Low Caffeine Group (≤200 mg/day): Individuals consuming caffeine within recommended levels (20-200 mg/day).
  Interventions: Other: Low Caffeine Consumption

INTERVENTIONS:
Other: High Caffeine Consumption — Individuals consuming 300 mg or more of caffeine daily, meeting DSM-5/ICD-10 criteria for caffeine dependence.
  Groups: High Caffeine Group (≥300 mg/day)
Other: Low Caffeine Consumption — Individuals consuming caffeine within recommended levels (20-200 mg/day).
  Groups: Low Caffeine Group (≤200 mg/day)

SUMMARY:
This study aims to evaluate the effects of caffeine dependence on hand reaction time and fine motor skills in university students. By comparing individuals with high and low daily caffeine intake, the research will assess whether excessive caffeine consumption is associated with impaired upper extremity performance. Reaction speed will be measured using the Nelson Hand Reaction Time Test, and manual dexterity will be assessed with the Purdue Pegboard Test.

DETAILED DESCRIPTION:
This observational study investigates the effects of caffeine dependence on hand reaction time and manual dexterity in young adults. Caffeine is a widely consumed psychoactive substance, and its excessive intake may influence motor and cognitive performance. University students aged 18 to 30 are recruited and divided into two groups based on daily caffeine consumption and diagnostic criteria from DSM-5/ICD-10: a high caffeine group (≥300 mg/day) and a low caffeine group (20-200 mg/day). Data are collected using the Caffeine Consumption Frequency Questionnaire and behavioral assessments conducted in a controlled laboratory environment. Hand reaction speed is measured with the Nelson Hand Reaction Time Test, while manual dexterity is assessed using the Purdue Pegboard Test. Sociodemographic data and caffeine consumption are gathered via online forms. The aim is to determine whether excessive caffeine intake is associated with changes in reaction time and fine motor skills. Statistical analyses include normality testing, group comparisons, and correlation analyses, with significance set at p<0.05. This study may provide new insights into the neuromotor effects of caffeine consumption in a university population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 30 years
* Currently enrolled university students

Exclusion Criteria:

* Neurological, vascular, orthopedic, acute or chronic conditions affecting hand function
* History of wrist surgery or visible hand deformity

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Healthy university students
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Nelson Reaction Time Test | Within the study duration (1 month)
  The Nelson Reaction Time Test assesses visual motor response time using a dropped ruler. The score is recorded in milliseconds, with lower scores indicating faster (better) reaction time. The test does not use a fixed scale with minimum or maximum values, but typical results range from approximately 100 ms to 300 ms depending on age and condition. Higher scores indicate slower (worse) reaction time.

SECONDARY OUTCOMES:
Purdue Pegboard Test | Within the study duration (1 month)
  The Purdue Pegboard Test evaluates manual dexterity and fine motor coordination. It consists of four subtests: right-hand, left-hand, both-hands, and assembly tasks. In the first three tasks, participants place as many pins as possible into holes on the board within 30 seconds using the specified hand(s). In the assembly task, participants assemble pegs, collars, and washers in sequence for 60 seconds. Scores are recorded as the number of pins or assembled parts placed correctly within the time limit. There is no fixed maximum score; however, higher scores indicate better manual dexterity and coordination.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided